CLINICAL TRIAL: NCT06308107
Title: Safety and Feasibility of Hyperkalemic Cardioplegia With Diazoxide in Cardiac Surgery (CPG-DZX) Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Magic That Matters (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00433127
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Stunning
MeSH Terms: conditions — Myocardial Stunning | interventions — Diazoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diazoxide (Experimental): IV Diazoxide as additive to hypothermic hyperkalemic cardioplegia.
  Interventions: Drug: IV Diazoxide

INTERVENTIONS:
Drug: IV Diazoxide — 500 micromoles added to one liter of cardioplegia

SUMMARY:
This study aims to confirm the safety and efficacy of diazoxide as an additive to hyperkalemic cardioplegia in patients undergoing cardiac surgery with cardiopulmonary bypass. The investigators hypothesize that diazoxide combined with hyperkalemic cardioplegia provides superior myocardial protection and reduced myocardial stunning compared with standard cardioplegia alone. Thirty patients will receive treatment. Safety will be assessed by comparing mean arterial blood pressure measurements, glucose levels and incidence of adverse events between the two groups. Efficacy will be assessed by comparing right and left ventricular function in pre-operative vs post-operative transesophageal echocardiograms, need for mechanical circulatory support, ease of separation from bypass and Vasoactive Inotrope Score (VIS) between the two groups. The information gained could pave the way for the use of Katp (Potassium-atp) channel openers to prevent stunning, improve patient outcomes, and reduce health care costs related to myocardial stunning that requires inotropic and mechanical support following cardiac surgery.

DETAILED DESCRIPTION:
This is a Phase I clinical trial. Thirty patients total will receive treatment (IV Diazoxide added to cardioplegia). Diazoxide will be added to the first dose of cardioplegia only. Subsequent doses of cardioplegia will not contain additives.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for cardiac surgery with cardiopulmonary bypass and cardioplegic arrest
* Patient scheduled for elective cardiac surgery
* If female participant of childbearing potential, she must agree to and be able to use a highly effective method of birth control (eg, barrier contraceptives, hormonal contraceptives, intrauterine devices, or sexual abstinence) continuously for six days post- diazoxide dose

Exclusion Criteria:

* Patient with Diabetes Mellitus on sulfonylurea medications
* Scheduled for left ventricular assist device (LVAD) or heart transplant
* Left ventricular ejection fraction < 30%
* Pre-operative placement or planned use of mechanical circulatory support during surgery
* Allergy to Thiazide and its derivatives
* History of gout
* Patient is pregnant or breastfeeding
* Patients with seizure disorders controlled by diphenylhydantoin
* Patients with a history of cold agglutinins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by mean change in blood pressure | From first dose of cardioplegia through 24 hours post operatively
  Mean blood pressure measurements in mmHg.
Safety as assessed by change in blood glucose levels | From first dose of cardioplegia through 48 hours post operatively
  Blood glucose levels in mg/dl.
Safety as assessed by incidence of adverse events | From first dose of cardioplegia through 7 days post operatively or discharge, whichever comes first
  Safety will be assessed by total number of adverse events.

SECONDARY OUTCOMES:
Efficacy as assessed by change in ejection fraction | Day of surgery (pre and post surgery)
  Comparison of right and left ventricular function (measured as a percentage) on pre and post operative Transesophageal echocardiograms
Efficacy as assessed by use of mechanical circulatory support | 48 hours post operatively
  Incidence of mechanical circulatory support use will be used in the assessment of efficacy.
Efficacy as assessed by change in Vasoactive Inotropic Score (VIS) | 0, 24, 48 and 72 hours post operatively
  Comparison of VIS Score with values from 0 to >45, with lower scores indicating medication efficacy (0e5, >5e15, >15e30, >30e45, and >45 points).
Efficacy as assessed by time to separate from Cardiopulmonary Bypass (CPB) | Day of surgery
  From time of first turn down of CPB to CPB end time measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lawton, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No